CLINICAL TRIAL: NCT03739190
Title: A 3-way Cross-over, Multi-centre Clinical Investigation to Evaluate the Performance Rate of Natural Rubber Latex Condoms of Varying Thickness in Healthy Monogamous Couples
Brief Title: A Clinical Investigation to Assess the Performance of Natural Rubber Latex Condoms in Couples
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 5005901
Record Dates: First submitted 2018-10-26; First posted 2018-11-13 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Control of Pregnancy; Prevention of Sexually Transmitted Infections

STUDY DESIGN:
Intervention Model Description: The condom types will be tested in a three-way cross-over design where couples will be randomised to use each of the three condom types in a defined order, according to the randomisation schedule.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each condom will be contained within an individual foil packet on which all branding will been masked. All the condom types will be masked in the same manner and identical boxes will be used for the test and comparator condoms A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Condom: Thin NRL Condom (Experimental): Following randomisation each couple will be given one set of 7 condoms as per randomisation schedule. Couples will return to the clinic site for collection of their next set of condoms on two additional occasions. Each couple will test a maximum of 21 condoms during their participation in the investigation.
  Interventions: Device: NRL Condom
- Reference condom A: Medium Thickness NRL Condom (Active Comparator)
  Interventions: Device: NRL Condom
- Reference condom B: Thick NRL Condom (Active Comparator)
  Interventions: Device: NRL Condom

INTERVENTIONS:
Device: NRL Condom — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to Subjects to be used during vaginal intercourse over a 4 week period, the assessment period. Couples will repeat the assessment period each of the 3 condom types.

SUMMARY:
This investigation is designed to evaluate the performance rate of a new natural rubber latex (NRL) male condom.

DETAILED DESCRIPTION:
In this clinical investigation, a new NRL male condom (test condom) will be evaluated against two marketed NRL male condoms of varying thickness (condom A and condom B). This clinical investigation will also evaluate the in-use tolerance of the test and the two reference condoms.

ELIGIBILITY:
Inclusion Criteria:

1. A male and a female subject aged: 18 - 60 years inclusive.
2. All subjects must be generally healthy and in a mutually monogamous heterosexual relationship - current relationship ≥ 3 months.
3. All couples must be sexually active, and agree to have penile-vaginal intercourse with a frequency sufficient to meet protocol requirements (a minimum of 5 coital acts over 4 weeks).
4. The female partner should use one other established highly effective form of non-barrier contraception, unless post-menopausal.
5. Couples must agree not to use drugs or non-investigational devices that can affect sexual performance e.g. medication/medical devices used to treat erectile dysfunction.

Exclusion Criteria:

1. Either partner is or becomes aware of an allergy or sensitivity to the ingredients of the test products, including the test or control condoms or any lubrication products provided.
2. Either partner has a pre-existing skin condition (severe eczema/psoriasis) or systemic allergic reactions or as confirmed by the subject and physical examination.
3. Either partner that needs to use condoms for a specific sexually transmitted infection (STI) protection e.g. discordance for Human Immunodeficiency Virus (HIV) or herpes.
4. Subjects that have previous or planned genital surgery, that in the opinion of the Investigator would consider the subject unsuitable to participate in the clinical investigation e.g. laser for abnormal smear.
5. Male partners that have known erectile or ejaculatory dysfunction.
6. Either partner that requires to use/is using medication or preparations that are applied topically to the genitalia area or intravaginally other than that supplied for the investigation.
7. A female partner that has been diagnosed with or treated for vaginal complaints (including vaginal dryness) in the previous 3 months which, in the opinion of the investigator, deems the partner unsuitable for the investigation.
8. Any participant who has clinical symptoms or signs of a sexually transmitted diseases (STD) or HIV/AIDS or has a previous history of high risk behaviour as judged by the investigator.
9. Female partner using medication which in the investigators opinion would affect vaginal mucosal secretion, such as Chlorpheniramine at any time in the 14 days (or 5 half-lives of the drug, whichever is longer) before first condom use.
10. A male partner with abnormal penile anatomy that would, in the opinion of the investigator, affect the ability to keep the condom in place during intercourse.
11. Either partner intends to continue to use antihistamines, anti-inflammatory drugs or pain killers for the duration of the investigation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 470 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Compared clinical failure rate of condom use between the test condom group and the reference condom A group | within 2 hours following each coital act for each condom use
  Number of clinical failure events, defined in ISO 29943-1:2017, will be reported by participants.
  Clinical failure rate is calculated as the number of condoms with at least 1 acute failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. A condom that experiences multiple clinical failure events only counts as a single clinical failure.

SECONDARY OUTCOMES:
Compared clinical failure rate of condom use between the test condom group and the reference condom B group | within 2 hours following each coital act for each condom use
  Number of clinical failure events, defined in ISO 29943-1:2017, will be reported by participants.
  Clinical failure rate is calculated as the number of condoms with at least 1 acute failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. A condom that experiences multiple clinical failure events only counts as a single clinical failure.
Compared clinical failure rate of condom use between the test condom group, the reference condom A group and reference condom B group | within 2 hours following each coital act for each condom use
  Number of clinical failure events, defined in ISO 29943-1:2017, will be reported by participants.
  Clinical failure rate is calculated as the number of condoms with at least 1 acute failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. A condom that experiences multiple clinical failure events only counts as a single clinical failure.
Incidence of treatment-emergent adverse events and adverse device effects, defined in MEDDEV 2.7/3 | 16 weeks
Subject's experience on the use of each type of condoms [Acceptability and Tolerability] | 16 weeks
  Acceptability and tolerability as assessed by subject perceived questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand